CLINICAL TRIAL: NCT05891067
Title: The Effectiveness of a Classroom-based Intervention Promoting Proscial Classroom Climate in Children
Brief Title: The Effectiveness of a Classroom-based Intervention Promoting a Prosocial Classroom Climate in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht University (Other)
Collaborators: KiVa B.V. (Unknown); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Amanda van Loon, Postdoc, Utrecht University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UtrechtU; 23-0082 (Other: Utrecht University)
Record Dates: First submitted 2023-04-28; First posted 2023-06-06 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: The design of the current study is a cluster Randomized Controlled Trial (RCT) with two conditions: the intervention condition and a waitlist control condition (TAU: treatment-as-usual). Schools are randomized into the intervention or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SterkWerk (Experimental): SterkWerk is a classroom-based approach (throughout the school year) for primary school groups 5-8 (children aged 8-12 years old) in which children are given specific roles to actively work on responsibility, ownership and prosocial behavior. SterkWerk consists of three main components: meaningful roles, classroom meeting and compliments.
  Interventions: Behavioral: SterkWerk
- Treatment-as-usual (Active Comparator): Schools in the control group do not receive the intervention (do not receive material or training), and function as normal (treatment-as-usual). Control schools are requested to not start any social-emotional program during the school year 2023/2024.
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: SterkWerk — Classroom-based intervention program
  Arms: SterkWerk
Behavioral: Treatment-as-usual — Active control group
  Other Names: TAU
  Arms: Treatment-as-usual

SUMMARY:
The purpose of this study is to investigate whether a classroom-based program promoting a prosocial classroom climate is more effective than treatment-as-usual (control condition).

DETAILED DESCRIPTION:
A positive, prosocial classroom climate is associated with improved social competence and academic achievement, as well as decreased internalizing and externalizing problems and antisocial behavior in children. It is expected that motivation to behave prosocially is needed to achieve a prosocial climate in the classroom, and that such motivation can be enhanced through three components of self-determination theory (SDT): competence, relatedness, and autonomy. The goal of this study is to examine the effectiveness of a classroom-based program based on SDT that aims to promote prosocial classroom climate, through a cluster Randomized Controlled Trial (RCT). SterkWerk is hypothesized to be more effective than treatment-as-usual (TAU) in creating more prosocial classrooms, through improving prosocial (intrinsic) motivation and behavior, social autonomy, social competence, and social relatedness.

The design of the current study is a cluster Randomized Controlled Trial (RCT) with two conditions: the intervention condition and a waitlist control condition (TAU: treatment-as-usual). Schools in the intervention condition receive the materials and training to implement the intervention in the school year 2023/2024. Schools in the control group do not receive the intervention (do not receive material or training), and function as normal (TAU). Control schools are requested to not start any social-emotional program during the school year 2023/2024.

ELIGIBILITY:
Inclusion Criteria:

* Primary school children of grades 5-8 (mostly aged between 8-12 years)
* Teachers and school leaders of participating schools (no age limit)

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3360 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in prosocial behavior as an injunctive form assessed with three items specifically developed for this study | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  It is a self-reported instrument rated on a 3-point scale from 1 (not true) to 3 (definitely true), measuring children's attitudes towards prosocial behavior that are on average held in the classroom. Higher scores reflect a higher injunctive norm of the group towards prosocial behavior.
Change in individual prosocial behavior assessed with four items based on the subscale prosocial behavior of the Strengths and Difficulties Questionnaire | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  The adapted SDQ subscale prosocial behavior is a self-reported instrument rated on a 4-point scale from 1 (never) to 4 (always). Higher scores reflect more prosocial behavior.
Change in prosocial relations in the classroom assessed with sociometric nominations | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  Children see a list with the names of all classmates and select the classmates that fit the question best according to them. Two items are used, assessing the child's prosocial behavior according to classmates. The number of received nominations is devided by the number of possible nominations, resulting in a proportion score for prosocial relations.
Change in cooperation and conflict in the classroom assessed with the Classroom Peer Context Questionnaire (CPCQ), subscales cooperation and conflict. | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  The CPCQ is a self-reported instrument. The cooperation subscale consists of four items assessing the extent to which children experience positive behavior. The conflict subscale consists of two items assessing the extent to which children experience negative behavior. The items are rated on a 4-point scale ranging from 1 (not true) to 4 (completely true). Higher scores on the cooperation subscale reflects more positive behavior, while for the conflict subscale it reflects more negative behavior.
Change in intrinsic (prosocial) motivation assessed with four items specifically developed for this study | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  This instrument is a self-reported instrument, rated on a 3-point scale ranging from 1 (not true) to 3 (definitely true). Higher scores reflect more intrinsic (prosocial) motivation.
Change in social competence assessed with five items based on the Rosenberg Self-Esteem Scale (RSES) | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  The adapted RSES is a self-reported istrument, rated on a 3-point scale ranging from 1 (not true) to 3 (definitely true). Higher scores reflect more social competence.
Change in social autonomy assessed with five items based on the School as a Caring Community Profile-II (SCCP-II) and the Child Development Project | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  It is a self-reported instrument, rated on a 4-point scale ranging from 1 (never) to 4 (always). Higher scores reflect more autonomy.
Change in social relatedness assessed with the Classroom Peer Context Questionnaire (CPCQ), subscales comfort and cohesion. | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  The CPCQ is a self-reported instrument. The comfort subscale consists of four items assessing the extent to which children feel at ease in the classroom. The cohesion subscale consists of two items assessing the extent to which the children in the classroom spend time together. The items are rated on a 4-point scale ranging from 1 (not true) to 4 (completely true). Higher scores on both subscales reflect more positive behavior.

SECONDARY OUTCOMES:
Change in school wellbeing assessed with seven items specifically developed for this study | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  This is a self-reported instrument. School belonging is measured with 7 items, rated on a 4-point scale ranging from 1 (never) to 4 (always). Higher scores reflect positive school wellbeing.
Change in school wellbeing assessed with one item specifically developed for this study | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  This is a self-reported instrument. School safety is measured with 1 item, rated on a 7-point scale ranging from 1 (very unsafe) to 7 (very safe). Higher scores reflect positive school wellbeing.
Change in social position (kindness, leadership, unkindness, popularity, best friends) assessed with sociometric nominations | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  Children see a list with the names of all classmates and select the classmates that fit the question best according to them. Five items are used, assessing the child's social position according to classmates. The number of received nominations is devided by the number of possible nominations, resulting in a proportion score for each social position (kindness, leadership, unkindness, popularity, best friends).
Change in bullying and bullying victimization assessed with the Olweus Bully-Victim Questionnaire (OB-VQ) | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  The OB-VQ is a self-reported instrument, consisting of items related to bullying, bullying victimization and the perceived behavior and attitudes of the teacher. Nine items related to bullying and victimization are rated on a 5-point Likert scale ranging from 1 (I did not bully / I was not bullied) to 5 (several times a week). Higher scores reflect more bullying and victimization.
Change in bullying and bullying victimization (where child is victimized) assessed with the Olweus Bully-Victim Questionnaire (OB-VQ) | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  The OB-VQ is a self-reported instrument, consisting of items related to bullying, bullying victimization and the perceived behavior and attitudes of the teacher. One item asks where the child is bullied. with answer options such as: in the halway, on the way to school, in the classroom (with the teacher present).
Change in bullying and bullying victimization assessed with the Olweus Bully-Victim Questionnaire (OB-VQ) | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  The OB-VQ is a self-reported instrument, consisting of items related to bullying, bullying victimization and the perceived behavior and attitudes of the teacher. Three items relate to the perceived behavior and attitude of the teacher. Higher scores reflect more negative attitudes/behavior of the teacher.
Change in bullying and bullying victimization assessed with sociometric nominations | T1 (baseline); T2 (mid-intervention) approximately 5 months after the start of the intervention; T3 (postintervention) approximately 10 months after the start of the intervention
  Regarding sociometric nominations,10 questions related to bullying victimization and one question related to bullying will be asked to children. Children see a list with the names of all classmates and select the classmates that fit the question best according to them. The number of received nominations is devided by the number of possible nominations, resulting in a proportion score for bullying.

OTHER OUTCOMES:
Child characteristics assessed with items specifically developed for this study | T1 (baseline)
  Child characteristics include age, gender, romantic attraction , grade, and ethnic identity (9 items).
Teacher characteristics assessed with items specifically developed for this study | T1 (baseline)
  Teacher characteristics include age, gender, years of experience (as a teacher in general, and as a teacher at the specific school) and experience with implementing social safety programs (10 items).
School characteristics assessed with items specifically developed for this study | T1 (baseline)
  School characteristics include location, number of participating grades and students in the classrooms, and years of experience with a social safety program (e.g., KiVa) (15 items).
Working elements (i.e., meaningful roles, weekly meetings and compliments) assessed with items specifically developed for this stuy | T2 (mid-intervention) approximately 5 months after the start of the intervention
  Children fill in questionnaires related to the three main components of the program: 1) meaningful roles (e.g., "How much did you like the role(s)" (12 items), 2) classroom meetings (e.g., "The weekly meetings were done independently by the class", 4 items), and 3) compliments (e.g., "I have received compliments from my classmates", 7 items). Higher scores reflect a more positive or greater adherence of the working elements.
Working elements (i.e., meaningful roles, weekly meetings and compliments) assessed with items specifically developed for this stuy | T3 (postintervention) approximately 10 months after the start of the intervention
  Teachers fill in questionnaires related to the three main components of the program: 1) meaningful roles (e.g., "Which roles were the most popular?", 9 items), 2) classroom meetings (e.g., "How often has a meeting been held?", 5 items), and 3) compliments (e.g., "How many times a week has attention been paid to the compliments?", 6 items). Higher scores reflect a more positive or greater adherence of the working elements.
Program integrity assessed with items specifically developed for this study | T2 (mid-intervention) approximately 5 months after the start of the intervention
  Teachers and school leaders fill in questionnaires related to the implementation of the program, divided into the domains training and material (e.g., "How often have you used the manual?", 9 items), child questionnaires (e.g., "Where there any questions that the children struggled with?", 2 items), time investment (e.g., "How did you feel about the time you had to implement the program properly?", 3 items), and global impression (e.g., "What is your general impression of the degree of success of the implementation of the program?", 6 items). Higher scores reflect a more positive or greater adherence of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Kaufman, dr., Principal Investigator — Utrecht University
Locations (1):
- Utrecht University, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be stored in a publicly available repository.
Supporting Information: Study Protocol
Time Frame: The data will become available after the completion of the program and data collection.
Access Criteria: The data will become publicly available
URL: http://dans.knaw.nl/en

REFERENCES:
- [Derived] van Loon AWG, Kaufman TML. The effectiveness of the Dutch Meaningful Roles program in children: a study protocol for a cluster randomized controlled study. BMC Public Health. 2023 Jul 27;23(1):1440. doi: 10.1186/s12889-023-16362-8. PMID 37501078